CLINICAL TRIAL: NCT03609463
Title: Promoting Weight Loss and Stress Reduction in Overweight and Obese Patients With Type 2 Diabetes: a Feasibility Study of a Combination of a Small Change and Well-Being Intervention
Brief Title: Promoting Weight Loss and Stress Reduction in Overweight and Obese Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiara Rafanelli (Other)
Responsible Party: Sponsor-Investigator, Chiara Rafanelli, Professor of Clinical Psychology, University of Bologna
Organization: University of Bologna (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PWLPWB-CVD
Record Dates: First submitted 2018-07-11; First posted 2018-08-01 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2; Overweight and Obesity
Keywords: diabetes; overweight; obesity; well-being; behavioral; small change; weight loss
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Diabetes Mellitus; Behavior; Weight Loss | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A researcher adequately trained in the administration of questionnaires and interviews, and blinded to the experimental allocation of patients, will carry out all the evaluations.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Well-being and small change (Experimental): Participants will be randomized to receive 4 individual 1-hour weekly sessions of the well-being intervention before starting the 12 individual 1-hour weekly sessions of the small change intervention in addition to the treatment as usual.
  Interventions: Behavioral: Small change intervention; Behavioral: Well-being intervention; Other: Treatment as usual
- Small change (Active Comparator): Participants will be randomized to receive 12 individual 1-hour weekly sessions of the small change intervention in addition to the treatment as usual.
  Interventions: Behavioral: Small change intervention; Other: Treatment as usual

INTERVENTIONS:
Behavioral: Small change intervention — The small change intervention is a behavioral intervention to help people gradually lose weight by making small changes in their lifestyle. At the beginning of the intervention participants will be met in person to be guided in setting an eating and a physical activity goal. Participants will be then contacted through the phone or met in person weekly for 3 months to check on their adherence to the selected goals and to discuss about facilitators and barriers to goal completion, in order to increase their motivation and problem solving skills. Every weekly contact will last about an hour and will be administered in an individual setting. At each contact selected goals can be revised, changed or another goal can be added based on levels of adherence.
Behavioral: Well-being intervention — The well-being intervention is a coaching intervention aimed at motivating people in making lifestyle changes by reducing levels of stress through the promotion of psychological well-being. It will consists in 4 weekly sessions to be held before starting the small change intervention. Each session will last about an hour and will be administered in an individual setting.
  Arms: Well-being and small change
Other: Treatment as usual — The treatment as usual includes any recommendation given to the participants by their physicians, including diet, physical activity, medication and glycemic control instructions.

SUMMARY:
This is a feasibility and acceptability study of a 16-month single-blind randomized controlled trial (RCT) designed to test the initial effectiveness of a well-being and small lifestyle changes intervention aimed at promoting weight loss and stress reduction in overweight and obese patients with type 2 diabetes. Primary goals of this study are to 1) evaluate study feasibility and patient acceptability, 2) develop a tailored protocol of a behavioral intervention for overweight or obese patients with type 2 diabetes that takes stress and well-being into consideration, 3) evaluate appropriateness of research procedures and measures, 4) examine effect size estimates of key outcomes to provide essential data to inform a larger efficacy trial, 5) determine whether clinically significant improvements occurred in any key outcomes.

DETAILED DESCRIPTION:
Overweight and obese patients with type 2 diabetes will be recruited at 2 different diabetes clinics. Physicians will screen every patient attending to each clinic during the enrollment period for the presence of main eligibility criteria. Those patients who appear to be eligible will be introduced to the study and referred to a researcher for a more in-depth screening evaluation. Eligible patients who are interested in participating in the study will be asked to sign the informed consent. Consecutive patients will be randomly assigned in a 1:1 ratio to an experimental group or a control group. During the first month, participants in the experimental group will receive a well-being promoting intervention in adjunction to the treatment as usual (TAU), while those in the control group will be asked to follow the TAU. In the following 3 months participants in both groups will receive the small change intervention in adjunction to the the TAU. All in person sessions of the intervention will take place in an office of both the 2 diabetes clinics involved. Data about psychological and clinical variables will be collected for each participant through questionnaires and interviews at baseline, at post-intervention, and at 6 and 12 months of follow-up. Participants' weight will be measured at each assessment point using a scale. Medical charts will be accessed to collect further data about physiological parameters, treatment received and medical history.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25;
* Age ≥ 18;
* Diagnosis of type 2 diabetes;
* Fluent English or Italian.

Exclusion Criteria:

* Inability to provide informed consent to participate in the study for any reason, including cognitive impairment and psychiatric illness;
* Presence of any medical condition that would make participation in the study difficult and/or unsafe;
* Presence of any medical condition associated with unintentional weight loss or gain;
* Presence of untreated, severe and/or recently diagnosed (≤ 6 months) mental illness and/or presence of a severe personality disorder;
* History of eating disorders and/or substance abuse;
* Use of drugs for weight loss;
* Participation in another weight loss program or in any other trial;
* Participation in an individual or group psychological intervention;
* Weight loss surgery within the year;
* Pregnant or are planning to become pregnant within the year
* Inability to control meal contents (e.g. institutionalized patients).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Feasibility (Recruitment) | Baseline
  Measured as the acceptance rate (total number of participants enrolled out of the total number of eligible candidates approached).
Feasibility (Retention) | Through study completion, intended to be 16 months
  Measured as drop-out rates (total number of participants who withdraw out of the total number enrolled).
Feasibility (Acceptability of Intervention) | Post-intervention, intended to be 4 months
  Measured as total number of sessions attended and number of weeks needed to complete the intervention. Semi-structured interviews will be conducted to estimate patients' satisfaction and provide data on optimal timing, dosing, and delivery.

SECONDARY OUTCOMES:
Change in Psychological Distress | Baseline, post-intervention (intended to be 4 months), 6 months post-intervention, 12 months post-intervention
  Measured by the Symptoms Questionnaire (SQ), a 92-item self-rating scale with yes/no responses (or true/false for some questions to avoid double-negative statements) divided into four domains: anxiety, depression, somatic, and anger-hostility.
  Each domain is further divided into two sub-scales: one sub-scale with 17 symptom questions and one sub-scale with 6 questions that are antonyms of some of the symptom questions in order to measure well-being.
  A response of yes/true for a symptom question gives 1 point, and a response of no/false for a well-being question gives 1 point for a score ranging from 0-17 for each symptom sub-scale and 0-6 for each well-being sub-scale, where a higher score indicates greater distress. If the well-being score is calculated separately the raw score can be subtracted from 6 for a score ranging from 0-6, where a higher score indicates greater well-being.
Change in Psychological Distress and Well-Being | Baseline, post-intervention (intended to be 4 months), 6 months post-intervention, 12 months post-intervention
  Measured by the Psychosocial Index (PSI), a 55-item self-rating scale divided into five domains:
  Sociodemographic and clinical data: 12 questions including routine medical and demographic information. Stress: 17 yes/no questions with a score from 0-17. A higher score indicates greater stress. Well-being: 6 yes/no questions with a score from 0-6. A higher score indicates greater psychological well-being. Psychological distress: 15 four-point questions from 0-3, with a total score from 0-45. A higher score indicates greater psychological distress. 4 questions referring to sleep may be scored separately. Abnormal illness behavior: 3 four-point questions from 0-3, with a total score from 0-9. A higher score indicates more severe abnormal illness behavior. Quality of life: 1 four-point question, with a score from 0 to 4. A higher score indicates a higher quality of life. Psychological well-being and quality of life scores can be summed for a global well-being score from 0-10.
Change in Psychological Well-Being | Baseline, post-intervention (intended to be 4 months), 6 months post-intervention, 12 months post-intervention
  Measured by the Psychological Well-Being scale (PWB), a 42-question self-rating scale for the assessment of 6 dimensions: self-acceptance, positive relations with others, autonomy, environmental mastery, purpose in life and personal growth. Each of the 42 six-point response questions are given a score from 1-6, with questions phrased in the negative reversed (e.g. 1 to 6, 6 to 1). The total score in each dimension ranges from 7-42, and all the dimensions scores are summed to give a final total ranging from 42-252, with higher scores indicating greater psychological well-being.
% Weight Change | Baseline, post-intervention (intended to be 4 months), 6 months post-intervention, 12 months post-intervention
  Measured in kg.

OTHER OUTCOMES:
Change in the Prevalence of Psychosomatic Syndromes | Baseline, post-intervention (intended to be 4 months), 6 months post-intervention, 12 months post-intervention
  Measured by the Diagnostic Criteria for Psychosomatic Research - Revised (DCPR-R), which uses a semi-structured interview of yes/no questions (DCPR-R SSI) to assess for the presence of 14 different psychosomatic syndromes. The prevalence will be reported as a within-population mean for each of the 14 syndromes described by the DCPR-R.
Change in Hemoglobin A1C | Baseline, post-intervention (intended to be 4 months), 6 months post-intervention, 12 months post-intervention
  Hemoglobin A1C levels will be obtained from patients' medical record.
Change in Abdominal Circumference | Baseline, post-intervention (intended to be 4 months), 6 months post-intervention, 12 months post-intervention
  Abdominal circumference will be measured in centimeters with a tape ruler.
Change in Physical Activity, Eating Habits, and Stress | Baseline, post-intervention (intended to be 4 months), 6 months post-intervention, 12 months post-intervention
  Measured by the GOSPEL questionnaire, a 32-item self-rating instrument for the assessment of physical activity levels, eating habits, and stress tailored to the dietary variation among Italian adults:
  Seven 4-point items regarding physical activity with a total score from 0 (least active) to 20 (most active).
  Ten 4-point items regarding diet based on frequency of consumption, with scores summed to obtain a Mediterranean diet score from 0 (worst) to 30 (best).
  Three 4-point items on eating habits summed for a score ranging from 0 (worst habits) to 9 (best habits).
  Diet and eating habits are summed to give a total diet score from 0 (worst) to 39 (best).
  Seven 4-point items regarding stress management summed for a total score from 0 (optimal management) to 21 (inadequate management).
  Four 4-point items on family risk behaviors with a score ranging from 0 (least risky) to 4 (most risky).
  One 4-point item on family support scored from 0 (least support) to 3 (most support).
Change in Food-Related Behaviors | Baseline, post-intervention (intended to be 4 months), 6 months post-intervention, 12 months post-intervention
  Measured by the Dutch Eating Behavior Questionnaire (DEB-Q), a 33-item self-rating instrument for the assessment of restrained (10 items), emotional (13 items), and external (10 items) eating behavior. Each item ranges from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the particular eating behavior, and thus a greater propensity to behavior associated with increased BMI. The mean score from each of the three sub-scales is reported.
Change in Motivation for Weight Loss | Baseline, post-intervention (intended to be 4 months), 6 months post-intervention, 12 months post-intervention
  Measured by the Goal Related Weight Questionnaire (GRWQ). The first section consists of 4 items and assesses the respondent's dream weight, happy weight, acceptable weight, and disappointed weight in kilograms. The respondent also writes the most important changes they hope to see following weight loss in one free-response question. The second section consists of 21 items asking the respondent to rate how they expect weight loss to impact various aspects of their psychosocial and health-related functioning, with each item scored from 1 (extremely negative) to 10 (extremely positive).
Change in Health-Related Quality of Life | Baseline, post-intervention (intended to be 4 months), 6 months post-intervention, 12 months post-intervention
  Measured by the 12-item Short Form Survey (SF-12), a 12-item self-rating scale for the assessment of physical and mental health comprising 8 domains: physical functioning, role-physical, bodily pain, general health, energy/fatigue, social functioning, role-emotional, mental health, and change in health. The weighted means of the 8 domains are calculated to develop two composite scores (Physical Health and Mental Health) ranging from 0 to 100, where 0 indicates the lowest level of health and 100 indicates the highest level of health.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Rafanelli, MD, PhD, Study Director — University of Bologna
Locations (2):
- Italy (2):
  - Struttura Semplice di Endocrinologia e Metabolismo, Ospedale Oglio Po, Casalmaggiore, Cremona
  - Servizio Endocrinologia e Diabetologia, Ospedale Bufalini, Cesena, Forlì-Cesena

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill JO. Can a small-changes approach help address the obesity epidemic? A report of the Joint Task Force of the American Society for Nutrition, Institute of Food Technologists, and International Food Information Council. Am J Clin Nutr. 2009 Feb;89(2):477-84. doi: 10.3945/ajcn.2008.26566. Epub 2008 Dec 16. PMID 19088151
- [Background] Phillips-Caesar EG, Winston G, Peterson JC, Wansink B, Devine CM, Kanna B, Michelin W, Wethington E, Wells M, Hollenberg J, Charlson ME. Small Changes and Lasting Effects (SCALE) Trial: the formation of a weight loss behavioral intervention using EVOLVE. Contemp Clin Trials. 2015 Mar;41:118-28. doi: 10.1016/j.cct.2015.01.003. Epub 2015 Jan 26. PMID 25633208
- [Background] Phillips EG, Wells MT, Winston G, Ramos R, Devine CM, Wethington E, Peterson JC, Wansink B, Charlson M. Innovative approaches to weight loss in a high-risk population: The small changes and lasting effects (SCALE) trial. Obesity (Silver Spring). 2017 May;25(5):833-841. doi: 10.1002/oby.21780. Epub 2017 Apr 5. PMID 28382755
- [Background] Geiker NRW, Astrup A, Hjorth MF, Sjodin A, Pijls L, Markus CR. Does stress influence sleep patterns, food intake, weight gain, abdominal obesity and weight loss interventions and vice versa? Obes Rev. 2018 Jan;19(1):81-97. doi: 10.1111/obr.12603. Epub 2017 Aug 28. PMID 28849612
- [Background] Fava GA. Well-Being Therapy: Current Indications and Emerging Perspectives. Psychother Psychosom. 2016;85(3):136-45. doi: 10.1159/000444114. Epub 2016 Apr 5. No abstract available. PMID 27043240
- [Background] Ryff CD. Psychological well-being revisited: advances in the science and practice of eudaimonia. Psychother Psychosom. 2014;83(1):10-28. doi: 10.1159/000353263. Epub 2013 Nov 19. PMID 24281296
- [Derived] Benasi G, Gostoli S, Zhu B, Offidani E, Artin MG, Gagliardi L, Rignanese G, Sassi G, Fava GA, Rafanelli C. Well-Being Therapy and Lifestyle Intervention in Type 2 Diabetes: A Pilot Randomized Controlled Trial. Psychosom Med. 2022 Nov-Dec 01;84(9):1041-1049. doi: 10.1097/PSY.0000000000001115. Epub 2022 Aug 2. PMID 36346956